CLINICAL TRIAL: NCT06039514
Title: Promoting Mental Health in Adolescents Through Mobile Apps: the Case of Eating Disorders.
Brief Title: Mobile App for Eating Disorders in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Principal Investigator, Gemma García-Soriano, Associate Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PID2021-124409OB-I00
Record Dates: First submitted 2023-09-04; First posted 2023-09-15 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Eating Disorders in Adolescence
Keywords: Maladaptive beliefs; Cognitive therapy; Eating Disorders; Mobile app; Adolescents; e-health
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Participants that meet the inclusion criteria will complete the web-based baseline assessment (pre), with questionnaires relating to maladaptive beliefs, emotional symptomatology, self-esteem, body satisfaction and eating symptomatology. After, experimental group will use the GGTCA-AD, and control group will use the GGNeutra for 14 days. Then, both groups will complete again the above-mentioned assessment (post use the app). Finally, all participants will complete the follow-up measures at one month.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GGTCA-AD mobile app (Experimental): The experimental group uses the GGTCA-AD module for 14 days after the first assessment.
  Interventions: Device: GGTCA-AD mobile app
- GGNeutra mobile app (Active Comparator): The control group uses GGNeutra for 14 days after the first assessment.
  Interventions: Device: GGNeutra mobile app

INTERVENTIONS:
Device: GGTCA-AD mobile app — The intervention will be done through an adaptation of the GGTCA app for teenagers: GGTCA-AD. This app is used to work on the dysfunctional beliefs that are associated with eating disorders. The app is made up of a series of levels comprising the topics that are normally worked on in cognitive behavior therapy (CBT) in relation to eating disorders. At each level, affirmations in the form of beliefs appear on the screen, and the person must accept them if they are functional, adaptive and positive; or reject them if they are dysfunctional, maladaptive and negative.
  Arms: GGTCA-AD mobile app
Device: GGNeutra mobile app — the control group will complete another module belonging to the GGTUDE digital platform. Specifically, this app is called GGNEUTRA, and the statements that compose it are totally independent of the target of the study. The operation is similar, sentences appear in the center of the screen, but in this case, the person must accept those sentences that are true, for example: "Madrid is the capital of Spain", by dragging it to the top of the screen; and reject those that are false, for example: "Tokyo is the capital of Spain", by dragging it to the bottom of the screen.
  Arms: GGNeutra mobile app

SUMMARY:
This study aims to evaluate the effectiveness of GGTCA-AD to decrease the maladaptive beliefs associated with eating disorders (ED) in non-clinical adolescent population. Specifically, a randomized controlled trial with parallel design and two groups (experimental and control) will be carried out in adolescents aged 13-15 years to assess the changes pre and post use of the app. It is expected that after the use of the GGTCA-AD app for 14 days, at the primary level, a: decrease in the degree of ascription to dysfunctional beliefs associated with ED; and at the secondary level: increase in body satisfaction and self-esteem; decrease in eating symptomatology; and no changes in emotional symptomatology. These results are also expected to be maintained in subsequent follow-up at 1 month.

DETAILED DESCRIPTION:
There is a digital platform called GGtude, which is composed of different modules, each of them aimed at working with different mental health problems. The goal is to provide an easy-to-use tool as a CBT complement to work on the self-dialogue that relates to the core beliefs associated with the psychological problem in particular. To achieve this target, a cognitive training exercise is performed: different sentences appear in the form of beliefs, and the person must identify and accept those beliefs that are functional, adaptive and positive, dragging them to the lower part of the screen; and reject those that are dysfunctional, maladaptive and negative dragging them to the upper part of the screen.

The GGTCA app is a module of GGtude that was developed to work on dysfunctional beliefs associated with eating disorders. Previous research showed that the app produced a statistically significant decrease of mean scores in maladaptive beliefs associated with ED and a statistically significant increase in self-esteem in adult population.

Furthermore, adolescence is a developmental stage vulnerable to the development of these disorders, so it's relevant to adapt the GGTCA application to the adolescent population (GGTCA-AD) and to evaluate its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

(1) ages between 13 and 16; (2) that the parents or guardians of the adolescents and the participants have signed the informed consent form; (3) have a dispositive with Internet access.

Exclusion Criteria:

(1) have inadequately answered control questions, for example "please check the option every day in this sentence".

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Change in the degree of ascription to dysfunctional beliefs associated with ED. | 15 days (after using the app) and one month later at follow-up.
  Score change in eating disorders maladaptive beliefs measured by the Eating Disorder Beliefs Questionnaire (EDBQ). It is composed of 32 items that examines core beliefs about weight, physical appearance and eating that are associated with eating disorders. Items are rated on an analog scale from 0 to 100, being 0 "I do not usually believe this at all" and 100 "I am usually completely convinced that this is true". Higher scores indicate the person has more maladaptive beliefs.

SECONDARY OUTCOMES:
Change in eating symptomatology. | 15 days (after using the app) and one month later at follow-up.
  Score change in eating symptoms measured by the Eating Disorder Examination Questionnaire (EDE-Q). It is a 36-item self-report questionnaire with 7-point Likert-type scale ranging from 0 (No day/ No time/ Not at all) to 6 (Every day/ Always/ Completely). It's composed of attitudinal and behavioral items, using for the present study only the attitudinal items (22 items). Higher scores indicate the person has greater presence of eating symptomatology.
Change in body satisfaction. | 15 days (after using the app) and one month later at follow-up.
  Score change in body satisfaction measured by the Body Appreciation Scale-2 (BAS-2). It is a single-factor questionnaire that evaluates body satisfaction with 10 items on a 5-point Likert scale (1 = Never; 5 = Always). Higher scores indicate the person has more body satisfaction.
Change in self-esteem. | 15 days (after using the app) and one month later at follow-up.
  Score change in self-report measures with The Single-Item Self-Esteem Scale (SISE; Robins et al., 2001). The person has to indicate how the statement "I have high self-esteem" describes him/her on a 9-point scale (1 = "Not very true for me" and 9 = "Very true for me"). Higher scores indicate the persona has more self-esteem.
Changes in emotional symptoms | 15 days (after using the app) and one month later at follow-up.
  No score change in depression and anxiety symptoms measured by The Patient Health Questionnaire for Depression and Anxiety (PH-4). It consists of 4 items, two for Anxiety and two for Depression, with a 4-point Likert scale (from 0 = "never" to 3 = "almost every day"). Higher scores indicate a greater presence of depression or anxiety symptoms.
Changes in perfectionism ans interpersonal distrust symptoms | 15 days (after using the app) and one month later at follow-up.
  Score change in perfectionism ans interpersonal distrust symptoms measured by the Eating Disorder Inventory (EDI-3), composed of 90 items with a 6-point Likert scale, where 0 = Never and 5 = Always. In this study only the interpersonal distrust and perfectionism factors are used, consisting of 7 and 6 items respectively. Higher scores indicate the person has greater presence of interpersonal distrust and perfectionism.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma García Soriano, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia/ Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Share all IPD that underlie results in a publication.
Time Frame: 3 months after the study is published.
Access Criteria: The variables analyzed will be included in the manuscript in which the RCT data are presented, and will be published on the institutional page of the applicants' university (https://roderic.uv.es/) up to 3 months after the article is published.
URL: http://roderic.uv.es/

REFERENCES:
- [Derived] Corberan M, Arnaez S, Saman Y, Pascual-Vera B, Garcia-Soriano G, Roncero M. Cognitive training via mobile app for addressing eating disorders' cognitions in adolescents: a randomized control trial protocol. BMC Psychol. 2024 May 14;12(1):268. doi: 10.1186/s40359-024-01772-z. PMID 38745260
- See also: Link to download the app from Google Play — https://play.google.com/store/apps/details?id=air.com.samuramu.gg.oc